CLINICAL TRIAL: NCT04033653
Title: Long-term Outcome Among Survivors of Sepsis in China Assessed by EQ-5D
Brief Title: Long-term Quality of Life Among Survivors of Sepsis in China Assessed by EQ-5D
Status: Completed | Type: Observational
Sponsor: Jianfeng Xie (Other)
Responsible Party: Sponsor-Investigator, Jianfeng Xie, Attending, Southeast University, China
Organization: Southeast University, China (Other)
Other Study IDs: sepsis long-term outcome
Record Dates: First submitted 2019-07-07; First posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sepsis is a common critical illness in Intensive Care Unit (ICU). With the continuous progress of severe medicine, the mortality rate of ICU hospitalization for sepsis has decreased, but the long-term prognosis is not satisfied. Due to the high long-term mortality, poor physical and mental health and cognitive impairment, the long-term quality of life decreases greatly, putting great burden on the family and society. Therefore, it is of great significance to understand the epidemiology and risk factors of the long-term prognosis of sepsis and find out how to improve the prognosis .

DETAILED DESCRIPTION:
Sepsis is a clinical syndrome in which the body's host response to uncontrolled infection leads to life-threatening organ dysfunction. In recent years, with the continuous improvement of the early diagnosis ability of sepsis, the deepening of the understanding of pathophysiology, and the continuous updating of treatment, the hospital mortality rate of sepsis has decreased significantly. However, studies have shown that the prevalence of sepsis is still increasing year by year, and the number of deaths due to sepsis is increasing. Sepsis is the main cause of death in ICU patients.

Although the mortality rate of patients with sepsis is significantly reduced, the increasing survival of patients with long-term outcome is not satisfied. All studies have shown that patients with sepsis have a high long-term mortality, and the long-term physiological, psychological, and cognitive function levels are reduced, which increases the economic burden and mental burden of the family and society. The increasing number of discharges has been considered a potential public health threat. In recent years, more and more researchers begin to pay attention to the long-term outcome of sepsis survivors. But compared with other acute or severe diseases, such as stroke, cancer, sepsis survivors has not been paid enough attention.

Therefore, all stages of treatment and rehabilitation of sepsis require extensive social attention. Continuous research and input are needed to explore predicting factors and effective interventions to improve the outcome and help patients and their families return to normal life,to reduce the social burden.

ELIGIBILITY:
Inclusion Criteria:

* survivors in the prior study (epidemiology survey of Chinese sepsis patients)

Exclusion Criteria:

* : patients who are unwilling to answer or lose their interviews

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: sepsis patients survived 90 days of oneset
Sampling Method: Probability Sample
Enrollment: 1368 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
2-year mortality | 2 year
  sepsis survivors will be followed up for 2-years
2-year readmission rate | 2 year
  sepsis survivors will be followed up for 2-years
mobility of sepsis survivors | 2 year
  one dimension of EQ-5D, which includes five dimensions and is used to evaluate the quaity of life of sepsis survivors. They are mobility， self-care，usual activities，discomfort or pain and depression or anxiety.
self-care of sepsis survivors | 2 year
  one dimension of EQ-5D, which includes five dimensions and is used to evaluate the quaity of life of sepsis survivors. They are mobility， self-care，usual activities，discomfort or pain and depression or anxiety.
usual activities of sepsis survivors | 2 year
  one dimension of EQ-5D, which includes five dimensions and is used to evaluate the quaity of life of sepsis survivors. They are mobility， self-care，usual activities，discomfort or pain and depression or anxiety.
discomfort or pain of sepsis survivors | 2 year
  one dimension of EQ-5D, which includes five dimensions and is used to evaluate the quaity of life of sepsis survivors. They are mobility， self-care，usual activities，discomfort or pain and depression or anxiety.
depression or anxiety of sepsis survivors | 2 year
  one dimension of EQ-5D, which includes five dimensions and is used to evaluate the quaity of life of sepsis survivors. They are mobility， self-care，usual activities，discomfort or pain and depression or anxiety.
the ability to judge and memory of sepsis survivors | 2 year
  It is scored by family or by yourself during telephone follow-up and is used to evaluate the quaity of life of sepsis survivors.

SECONDARY OUTCOMES:
influencing factors | 2 year
  explore the relationship between the outcome of sepsis survivors and clinical characteristics.The clinical characteristics is collected from Clinical case system,to explore their relationship with two-year survival, two-year quality of life of sepsis survivors.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yi, Ph.D., Study Director — Zhongda Hospital
Locations (1):
- Zhongda hospital, Southeast University, Nanjing, Jiangsu, China